CLINICAL TRIAL: NCT00875446
Title: A Single and Repeat Dose Escalation Study of the Safety, Pharmacokinetics and Pharmacodynamics of GSK1223249 in ALS Patients
Brief Title: First Time in Human Study of GSK1223249 in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 111330
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — ozanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects receiving GSK1223249 (Experimental): Eligible subjects will receive sequential dose of intravenous infusion of GSK1223249 with a starting dose of 0.01 milligram per kilogram followed by 0.1, 0.5,
  1, 2.5, 5, 7.5, and 15 milligrams per kilograms.
  Interventions: Drug: GSK1223249
- Subjects receiving placebo (Placebo Comparator): Eligible subjects will receive intravenous infusion of placebo.
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: PLACEBO — Placebo
  Arms: Subjects receiving placebo
Drug: GSK1223249 — I.V Infusion
  Arms: Subjects receiving GSK1223249

SUMMARY:
The drug being tested in this study is GSK1223249. It is being developed by GlaxoSmithKline to treat symptoms in patients with Amyotrophic Lateral Sclerosis (ALS).

The drug works by inhibiting the protein that prevents nerve growth.

This will be the first time the drug will be given to man. The trial is expected to involve approximately 76 patients. The study objective is to investigate the tolerability, safety and the way the body handles GSK1223249 after a range of single doses or repeat dose escalation in patients with ALS.

DETAILED DESCRIPTION:
This is the first-time-in-human (FTIH) phase I/IIa study of GSK1223249, a humanised monoclonal antibody against Nogo-A, a neurite outgrowth inhibitor hypothesised to be involved in the pathophysiology of amyotrophic lateral sclerosis (ALS) and some other neurodegenerative disorders. This study will be a randomized, placebo-controlled, double-blind, sequential dose escalation, 2-part fusion protocol. Approximately 76 patients with ALS will be enrolled. In Part 1, single escalating intravenous (i.v.) doses of GSK1223249 are planned to be evaluated in 5 sequential patient cohorts (2 placebo and 6 active in each cohort) to determine single dose safety and pharmacokinetics (PK). Part 2 will also be of a sequential dose escalating design, but patients in each of the planned 3 cohorts (3 placebo, 9 active in each cohort) will receive 2 repeat i.v. doses approximately 4 weeks apart where, safety and PK will also be evaluated. In two cohorts in Part 1 and all cohorts in Part 2, blood samples and skeletal muscle biopsies will be taken from patients before and at the end of treatment to demonstrate whether or not GSK1223249 binds to its target and produces any measurable pharmacodynamic effect. Patients in both parts will receive their first dose in a hospital-based unit where they will be monitored for at least 24 hours post-dose before being discharged to be followed on an out-patient basis. In each cohort in part 1, the first four subjects will be dosed in a staggered manner such that only one will receive the dose in any 24 hours. Dosing of the first four subjects in the first cohort of part 2 will also be staggered in a similar manner.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of familial or sporadic ALS, defined as meeting the possible, laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS according to the revised World Federation of Neurology El Escorial criteria [Rix Brooks 2000].
* Onset of muscle weakness within 60 months of study entry.
* Patients who have low Slow Inspiratory Vital Capacity (SVC) below that what is predicted for age and sex can be included into the study at the discretion of the investigator as long as they are NOT respiratory insufficient.
* If on any medication (including riluzole), these must have been stable within the previous one month. (See also 'Concomitant Medications' - Section 8).
* Age 18 - 80 years inclusive.
* Male or Female of non-childbearing potential (NCBP) defined as follows:

Pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and oestradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 7.1.1, if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

* Male subjects must agree to use one of the contraception methods listed in Section 7.1.2. This criterion must be followed from the time of the first dose of study medication until the last follow-up visit.
* QTcB < 500 msec or uncorrected QT <600msec (machine or manual overread). If subject has bundle branch block then criteria is QTcB < 530 msec.
* A Body Mass Index that at the discretion of the investigator is acceptable for inclusion into the study.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Patients with other neuromuscular disorders (in addition to their ALS diagnosis), unless the investigator determines that such additional disorder will not affect safety or other measures in this study.
* Patients with evidence of dementia or psychiatric illness which, in the investigator's opinion, is likely to prevent them from a full understanding of and/or compliance with the study requirements and procedures.
* Patients with abnormalities detected during the screening evaluations which, in the investigator's medical judgement, are sufficiently significant to exclude them from participation in the study.
* Patients who have participated in a clinical trial involving receipt of a biopharmaceutical product within 6 months prior to the first dosing day.
* Exposure to more than four new investigational products within 12 months prior to the first dosing day.
* The subject has a positive drugs of abuse test at the screening or pre dose visit. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates and benzodiazepines. Subjects who are on any of these drugs by prescription for medical reasons may be considered by the investigator for inclusion if they fulfil other entry criteria.
* The subject has a positive alcohol test at the pre-dose visit. History of regular excessive alcohol consumption within 6 months of the study defined as:
* For European sites: an average weekly intake of > 28 units for males or >21 units for females. One unit is equivalent to 8g of alcohol: a half-pint (~240mL) of beer, 1 glass (125mL) of wine or 1 (25mL) measure of spirits.
* For North American sites: an average weekly intake of >21 drinks for males or >14 drinks for women. One drink is equivalent to 12 g alcohol: 12 ounces (360mL) of beer, 5 ounces (150mL) of wine or 1.5 ounces (45mL) of 80 proof distilled spirits.
* History of sensitivity to GSK1223249, or components thereof, or a history of drugs or other allergies that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Females of childbearing potential, pregnant females as determined by positive serum or urine beta hCG test at screening or prior to dosing, or lactating females.
* Patients who have received any type of vaccination in the last 3 weeks before study drug administration.
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subjects who will undergo muscle biopsies (cohorts 3-optional 5, 6, 7 and 8 will not be eligible for inclusion, if any of the following criteria apply:

Patients with wasted deltoids (MRC score ≤ 2) and patients with normal deltoids (MRC score 5).

Patients who cannot achieve normal coagulation in the peri-operative period and those who may otherwise be at higher risk of bleeding complications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-05-13 (Actual); Primary Completion 2011-09-09 (Actual); Study Completion 2011-09-09 (Actual)

PRIMARY OUTCOMES:
Adverse events, vital signs, standard physical examination, ECG and standard clinical laboratory tests (haematology and biochemistry). Evaluation of safety will include any adverse effects on Immunogenicity, ALSFRS-R, SVC, Muscle Strength and MUNE. | 12-16 Weeks

SECONDARY OUTCOMES:
GSK1223249: Single dose PK (Part 1): AUC(0-∞), AUC(0-t), AUC(0-Week 4), %AUCex, Cmax, tlast, CL, Vss, MRT, λz and t½.Repeat dose PK (Part 2): GSK1223249 AUC(0-Week 4), Cmax and after the second dose, AUC(0-t), AUC(0-∞),λz and t½. | 12-16 Weeks
Presence of antibodies to GSK1223249 will be assessed in serum samples using immuno-electrochemiluminescent assay. | At least 16 weeks
ALSFRS-R scores, Manual Muscle Strength test and Slow Inspirational Vital Capacity (SVC) | 12-16Weeks
Motor Unit Number Estimation (MUNE) | 12-16 Weeks
Muscle biopsies for protein analysis, Immunohistochemistry (IHC), Transcriptomics. Blood for protein analysis and other biomarkers. | At least 16 weeks
Relationships between PK of GSK1223249 and relevant pharmacological endpoints | At least 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (6):
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Columbus, Ohio
- GSK Investigational Site, Paris, France
- GSK Investigational Site, Verona, Veneto, Italy
- United Kingdom (3):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London

REFERENCES:
- [Derived] Meininger V, Pradat PF, Corse A, Al-Sarraj S, Rix Brooks B, Caress JB, Cudkowicz M, Kolb SJ, Lange D, Leigh PN, Meyer T, Milleri S, Morrison KE, Orrell RW, Peters G, Rothstein JD, Shefner J, Lavrov A, Williams N, Overend P, Price J, Bates S, Bullman J, Krull D, Berges A, Abila B, Meno-Tetang G, Wurthner J. Safety, pharmacokinetic, and functional effects of the nogo-a monoclonal antibody in amyotrophic lateral sclerosis: a randomized, first-in-human clinical trial. PLoS One. 2014 May 19;9(5):e97803. doi: 10.1371/journal.pone.0097803. eCollection 2014. PMID 24841795
- See also: Results for study 111330 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111330?search=study&study_ids=111330#rs